CLINICAL TRIAL: NCT05144867
Title: Stereotactic Radiosurgery vs Whole Brain Radiotherapy in Breast Cancer With Brain Oligometastasis- A Randomised Controlled Phase 3 Trial
Brief Title: Stereotactic Radiosurgery vs Whole Brain Radiotherapy in Breast Cancer With Brain Oligometastasis
Acronym: SRSvsWBRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Budhi Singh Yadav, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK/7784/Study/249
Record Dates: First submitted 2021-11-02; First posted 2021-12-03 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Brain Metastases, Adult; Stereotactic Radiosurgery; Whole Brain Radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): The WBRT dosage schedule will be 30 Gy in 10 fractions over 2 weeks. For Arm 1, Treatment planning is to be done using CT simulation or conventional simulation (fluoroscopy). Simple beam arrangements, such as parallel opposed beams, will be favoured wherever possible.
  Interventions: Radiation: Stereotactic Radiosurgery
- Arm 2 (Experimental): Metastases with a maximum diameter of up to 2 cm will be treated with doses of 22 to 25 Gy and those larger than 2 cm will be treated with doses of 18 to 20 Gy.
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — All patients to undergo planning CT simulation with 1mm slice thickness. For all lesions, the gross tumor volume (GTV) will be defined as the visible tumor on CT and/or MRI imaging. A Planning Target Volume (PTV) margin of 2-5 mm will be added. Organs at risk visible in the planning CT scan will be contoured. The doses will be prescribed to approximately 100% isodose level and 95% of the PTV should receive 95% of the prescription dose. Metastases with a maximum diameter of up to 2 cm will be treated with doses of 22 to 25 Gy and those larger than 2 cm will be treated with doses of 18 to 20 Gy.

SUMMARY:
This trial aims to assess the impact of SRS on overall survival, PFS, radiation toxicity and quality of life as compared to WBRT in oligometastatic brain disease in breast cancer patients. Total 98 patients with breast cancer with brain oligo-metastases will be included. The WBRT dosage schedule will be 30 Gy in 10 fractions over 2 weeks. For tumors with 2cm, SRS dose of 22 to 25 Gy will be delivered and tumor larger than 2 cm will be treated with doses of 18 to 20 Gy.

DETAILED DESCRIPTION:
AIMS AND OBJECTIVES To assess the impact of SRS on overall survival, brain tumour recurrence and radiation toxicity with oligometastatic brain metastasis as compared to patients who receive WBRT.

Primary End Point: Overall Survival (OS) Secondary End Points: Progression Free Survival (PFS) Toxic Effects of Radiation Quality of Life DETAILED RESEARCH METHODOLOGY Study Setting: Department of Radiotherapy and Oncology, Post Graduate Institute of Medical Education and Research, Chandigarh Study Design: Prospective hospital based study

Inclusion criteria:

* Age >=18 years
* Willing to provide informed consent
* Histologically confirmed malignancy with metastatic disease detected on imaging.
* ECOG performance status 0-1
* 1 to 5 brain metastases, each with a maximum diameter of no more than 3.5 cm on contrast enhanced magnetic resonance imaging(MRI) scans.

Exclusion criteria

* Serious medical comorbidities
* ECOG >= 2
* Prior Brain Radiotherapy
* >5 brain metastasis
* Maximum diameter >4cm on MRI

Randomisation and Treatment:

Prior to randomization, a complete history and physical examination by the treating radiation oncologist will be done. Histologically confirmation of malignancy is required, with metastatic disease detected on imaging. Prior to randomization, the patients will be stratified based on number of brain metastases (single vs 2-3), extent of extracranial disease (active vs stable). Extracranial disease will be considered to be stable when the tumor had been clinically controlled for 6 months or longer prior to the detection of brain metastases. After informed consent, eligible patients will be randomised in two arms.

Arm 1:

The WBRT dosage schedule will be 30 Gy in 10 fractions over 2 weeks. For Arm 1, Treatment planning is to be done using CT simulation or conventional simulation (fluoroscopy). Simple beam arrangements, such as parallel opposed beams, will be favoured wherever possible.

Arm 2:

All patients in Arm 2 will undergo planning CT simulation with 1mm slice thickness. For all lesions, the gross tumor volume (GTV) will be defined as the visible tumor on CT and/or MRI imaging. A Planning Target Volume (PTV) margin of 2-5 mm will be added. Organs at risk visible in the planning CT scan will be contoured. The doses will be prescribed to approximately 100% isodose level and 95% of the PTV should receive 95% of the prescription dose. Metastases with a maximum diameter of up to 2 cm will be treated with doses of 22 to 25 Gy and those larger than 2 cm will be treated with doses of 18 to 20 Gy.

Follow up:

Clinical evaluations and MRI scans will be done 1 and 3 months after treatment and every 3 months thereafter. In cases in which a recurrence will be detected, further treatment can be administered. The size of the treated lesions will be measured in 3 dimensions, and this size, the development of new brain metastases, and the development of leukoencephalopathy associated with radiological findings (according to the National Cancer Institute's Common Toxicity Criteria version 4.0319) will be scored based on serial MRI scans. Overall survival will be measured as time until death from any cause, and progression-free survival as time to either progression or death, whichever occurs first. Lesion response will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee20. At each visit, functional status and neurologic toxic effects will be scored. Systemic functional status will be evaluated by using the KPS score. Neurologic function will be evaluated according to the criteria listed21.

Statistical analysis:

This study will aim to detect an improvement in overall survival. The study will therefore be designed with 80% power. It is estimated that the median survival of the control group after randomization in this study will be 9 months. In order to detect a 6-month improvement in median survival from 9 months to 15 months with SRS, a total of 93 patients will be needed. Assuming a 5% rate of loss to follow up, a total of 98 patients will be accrued. The study projects accrual over 48 months with 12 months of additional follow-up. Survival will be calculated using the Kaplan-Meier method with differences compared using the stratified log-rank test. A Cox multivariable regression analysis will be used to determine baseline factors predictive of survival. Differences in rates of grade 2 or higher toxicity between groups will be tested using the Fisher's Exact Test. Differences in progression free survival will be tested using the stratified log-rank test.

Novelty of study: This trial aims to assess the impact of SRS on overall survival, PFS, radiation toxicity and quality of life as compared to WBRT in oligometastatic brain disease in breast cancer patients. It may lead to better understanding of role of SRS in oligometastatic paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Willing to provide informed consent
* Histologically confirmed malignancy with metastatic disease detected on imaging.
* ECOG performance status 0-1
* 1 to 3 brain metastases, each with a maximum diameter of no more than 3 cm on contrast enhanced magnetic resonance imaging(MRI) scans

Exclusion Criteria:

* Serious medical comorbidities
* ECOG >= 2
* Prior Brain Radiotherapy
* >3 brain metastasis
* Maximum diameter >4cm on MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  From date of randomization till death due to breast cancer

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 1 year
  From completion of radiotherapy treatment to intracranial progression of disease on MRI/CT scan as per the RECIST criteria which is >20% increase(>5mm absolute increase) in the the sum of the longest diameters in comparison with the smallest sum of the longest diameters recorded since treatment started.
Quality of Life - KPS | Base line and 6 months
  At each visit, functional status and neurologic toxic effects will be scored. Systemic functional status will be evaluated by using the KPS score. KPS will be scored 80-100 if the patient is able to carry on normal activity and to work without special care. A score of 50-70 will indicate patient is unable to work; live at home and care for most personnel needs; varying amount of assistance required. A score of 10-30 indicate that unable to care for self; requires equivalent of hospital or institutional care; disease may be progressing rapidly. A score of 0 means patient is dead. Neurologic function will be evaluated according to the MINI MENTAL STATE EXAMINATION. Patients will be scored for each question from 0-30. Degree of impairment will be graded as severe if the score is 0-10, moderate if the score is 10-20, mild between 20-25 and questionable significant if the score is 25-30.
Quality of life - MINI MENTAL STATE | Base line and 6 months
  Neurologic function will be evaluated according to the MINI MENTAL STATE EXAMINATION. Patients will be asked a set of questions( for example what is the year? season? date? day? month?; where are we now? state? county? town? city? hospital?; spell WORLD back word or count D-L-R-O-W or count back word from 100 by seven- 93, 86, 79, 72, 65). Score 1 point for each correct response with in each question will be given so that a score from 0-30 is recorded. Degree of impairment will be graded as severe if the score is 0-10, moderate if the score is 10-20, mild between 20-25 and questionable significant if the score is 25-30.

CONTACTS AND LOCATIONS:
Overall Officials: Budhi Singh Yadav, MD, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- Budhi Singh Yadav, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta A, Yadav BS, Ballari N, et al. LINAC-based stereotactic radiosurgery/radiotherapy for brain metastases in patients with breast cancer. Journal of Radiotherapy in Practice , Volume 21 , Issue 3 , September 2022 , pp. 351 - 359 DOI: https://doi.org/10.1017/S1460396921000029[Opens in a new window]
- [Derived] Yadav BS, Vias P, Robert N, Gade VKV, Kajla A. Whole Brain Radiotherapy Versus Stereotactic Radiosurgery in Breast Cancer Patients With Brain Metastases-A Phase 3 Open Label Randomized Study. Asia Pac J Clin Oncol. 2025 Sep 22. doi: 10.1111/ajco.70029. Online ahead of print. PMID 40983872